CLINICAL TRIAL: NCT06031220
Title: Response of Pulmonary Functions to Deep Breathing Exercise in Twin Pregnancy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Badr University (Other)
Responsible Party: Principal Investigator, Noha Ahmed Fouad Abd-Elrahman, lecturer of physical therapy for women health, Badr University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: P.T.REC/012/004052
Record Dates: First submitted 2023-09-03; First posted 2023-09-11 (Actual); Last update posted 2023-11-22 (Actual); Status verified 2023-11

CONDITIONS: Pregnancy Related

STUDY DESIGN:
Who Masked: Participant
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- study group (Experimental): 30 women with twin pregnancy during the third trimester at 27th weeks gestation will make deep breathing exercise inform of diaphragmatic and costal breathing 3times a day for 15 repetitions each exercise for 9 weeks, pulmonary function test will be applied at 27th week gestation and at 36th weeks gestation.
  Interventions: Other: deep breathing exercise inform of diaphragmatic and costal breathing
- control group (No Intervention): 30 women with twin pregnancy during the third trimester at 27th weeks gestation will not receive any special treatment and will be assessed with pulmonary function test at 27th week gestation and at 36th weeks gestation.

INTERVENTIONS:
Other: deep breathing exercise inform of diaphragmatic and costal breathing — deep breathing exercise inform of diaphragmatic and costal breathing 3times a day for 15 repetitions each exercise for 9 weeks,
  Arms: study group

SUMMARY:
this study is to investigate the response of pulmonary function to deep breathing exercise in twin pregnancy

DETAILED DESCRIPTION:
Physiological changes during pregnancy impose numerous changes on the respiratory system that can affect the health of both mother and foetus. Regarding the importance of the normal breathing in the health of mother and foetus.

Many investigators have studied pulmonary function tests during normal pregnancy, most of them found a significant decrease in pulmonary function test parameters during all pregnancy trimesters. Others showed that the PFTs parameters are normal in the first trimester but there was significant decrease in them in the second and third trimesters, or in the third trimester only.

Study Design: Randomized control trial Sixty twin pregnant women during the third trimester i (27th weeks gestation),aged 25 to 35 years old and body mass index was ≥ 30 kg/m², will participate in this study. They will be assigned into two equal groups; control group and study group ( study group only will make deep breathing exercise inform of diaphragmatic and costal breathing 3times a day for 15 repetitions each exercise for 9 weeks, pulmonary function test will be applied for both groups at 27th week gestation and at 36th weeks gestation.

ELIGIBILITY:
Inclusion Criteria:

* All pregnant women will be in 27th week gestation
* They will be recruited from Soaad kafafy university hospital
* Their age between 25-35 years old
* Their BMI ≥30Kg/m2

Exclusion Criteria:

* Pregnant women with any pulmonary disorders before pregnancy
* Women suffering from any physical or mental disorders.
* Pregnant women with gestational diabetes
* Pregnant women with gestational hypertension
* Pregnant women with asthma

Ages: 25 Years to 35 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 60 (Actual)
Dates: Start 2022-10-01 (Actual); Primary Completion 2023-05-30 (Actual); Study Completion 2023-06-05 (Actual)

PRIMARY OUTCOMES:
forced vital capacity (FVC) | FVC will be applied at 27th week gestation and at 36th weeks gestation (3 months)
  inspiratory reserve volume + tidal volume+ expiratory reserve volume
Forced Expiratory Volume in 1 Sec (FEV1) | FEV1 will be applied at 27th week gestation and at 36th weeks gestation (3 months)
  Pulmonary Function Tests: (Forced Expiratory Volume in 1 Sec)
FEV1/FVC | FEV1/FVC will be applied at 27th week gestation and at 36th weeks gestation (3 months)
  ratio between Forced Expiratory Volume in 1 Sec (FEV1) and forced vital capacity (FVC)

CONTACTS AND LOCATIONS:
Overall Officials: Radwa S Mahmoud, PhD, Study Chair — Ass. Prof. Dept of PT for pediatrics, Faculty of PT, Cairo University and BUC; Shimaa HA roshdy, PhD, Study Chair — Lecturer of PT Dept of PT for cardiopulmonary and geriatric, Faculty of PT, MUST; Ayman A Elsallamy, PhD, Study Chair — Lecturer of obstetrics and gynecology, Ob/ GYN dept MUST; Doaa S Mohamed El-sayed, PhD, Study Chair — Lecturer of PT, Dept. of PT for women's health, Faculty of PT, BUC; Mina AG Elias, PhD, Study Chair — Lecturer of PT, Dept. of PT for internal medicine and geriatric, Faculty of PT, BUC; Noha A Fouad, PhD, Principal Investigator — Lecturer of PT, Dept. of PT for women's health, Faculty of PT, BUC
Locations (1):
- Soaad kafafy university hospital, Giza, Egypt